CLINICAL TRIAL: NCT01420393
Title: A Randomized Ablation-based Atrial Fibrillation Rhythm Control Versus Rate Control Trial in Patients With Heart Failure and High Burden Atrial Fibrillation
Brief Title: Rhythm Control - Catheter Ablation With or Without Anti-arrhythmic Drug Control of Maintaining Sinus Rhythm Versus Rate Control With Medical Therapy and/or Atrio-ventricular Junction Ablation and Pacemaker Treatment for Atrial Fibrillation
Acronym: RAFT-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 231888
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Heart Failure; Atrial Fibrillation
Keywords: Heart Failure; Atrial Fibrillation; Catheter Ablation; Anti-arrhythmic Medications; Cardiovascular Mortality
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation | interventions — Catheter Ablation; Heart Rate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rhythm Control (Active Comparator): Patients randomized to catheter ablation-based AF rhythm control group will receive optimal Heart Failure therapy and one or more aggressive catheter ablation, which include PV antral ablation and LA substrate ablation with or without adjunctive antiarrhythmic drug.
  Interventions: Procedure: Rhythm control
- Rate Control (Active Comparator): Patients in the rate control group will receive optimal Heart Failure therapy and rate control measures to achieve a resting HR < 80 bpm and 6-minute walk HR < 110 bpm.
  Interventions: Other: Rate Control

INTERVENTIONS:
Procedure: Rhythm control — Patients randomized to catheter ablation-based AF rhythm control group will receive optimal HF therapy and one or more aggressive catheter ablation, which include PV antral ablation and LA substrate ablation with or without adjunctive antiarrhythmic drug
  Other Names: Catheter ablation
  Arms: Rhythm Control
Other: Rate Control — Patients in the rate control group will receive optimal HF therapy and rate control measures to achieve a resting HR < 80 bpm and 6-minute walk HR < 110 bpm.
  Other Names: Standard medical therapy
  Arms: Rate Control

SUMMARY:
Atrial fibrillation and heart failure are two common heart conditions that are associated with an increase in death and suffering. When both of these two conditions occur in a patient the patient's prognosis is poor. These patients have poor life quality and are frequently admitted to the hospital. The treatment of atrial fibrillation in heart failure patients is extremely challenging. Two options for managing the atrial fibrillation are permitting the atrial fibrillation to continue but controlling the heart rate, or to convert the atrial fibrillation rhythm back to normal and try to maintain the heart in sinus rhythm. Until now, the method to keep the patient in normal sinus rhythm is with antiarrhythmic drugs. Studies using antiarrhythmic drugs to control the rhythm failed to show any survival benefit when compared with permitting the patient to be in atrial fibrillation. In the last few years, new development in techniques and technologies now enable catheter ablation (cauterization of tissue in the heart with a catheter) to be a successful treatment in abolishing atrial fibrillation and that this approach is better than antiarrhythmic drug to control the rhythm. However, there has not been any long-term study to determine whether catheter ablation to abolish atrial fibrillation in heart failure patients would reduce mortality or admissions for heart failure.

This study is to compare the effect of catheter ablation-based atrial fibrillation rhythm control to rate control in patients with heart failure and high burden atrial fibrillation on the composite endpoint of all-cause mortality and heart failure events defined as an admission to a healthcare facility for > 24 hours or clinically significant worsening heart failure leading to an intervention (defined as treatment in an emergency department, a same-day access clinic, or an infusion centre) or unscheduled visits to a healthcare provider for administration of an intravenous diuretic and an increase in chronic heart failure therapy. This study may have a dramatic impact on the way the investigators manage these patients with atrial fibrillation and heart failure and may improve the outlook and well being of these patients.

DETAILED DESCRIPTION:
Substudy_ In a subset of patients, following informed consent, additional data collection will include annual NT-proBNP/BNP measurements, Echocardiogram baseline and annually and 14 Day ECG Continuous Monitoring at six month intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with one of the following AF categories and at least one ECG documentation of AF

   * High burden Paroxysmal defined as ≥ 4 episodes of AF in the last 6 months, and at least one episode > 6 hours (and no episode requiring cardioversion and no episode > 7 days)
   * Persistent AF (1) defined as ≥ 4 episodes of AF in the last 6 months, and at least one episode > 6 hours, and at least one AF episode less than 7 days but requires cardioversion. No AF episodes are > 7 days
   * Persistent AF (2) as defined by at least one episode of AF > 7 days but not > 1 year
   * Long term persistent AF defined as an AF episode, at least one year in length and no episodes > 3 years
2. Optimal therapy for heart failure of at least 6 weeks (according to 2009 ACCF/AHA class 1 recommendations).
3. HF with NYHA class II or III symptoms with either impaired LV function (LVEF ≤ 45%) as determined by EF assessment within the previous 12 months or preserved LV function (LVEF > 45%) determined by by EF assessment within the previous 12 months
4. NT-pro BNP measures:

   A) Patient has been hospitalized for Heart Failure* in the past 9 months, has been discharged AND:

   i- Is presently in Normal Sinus Rhythm and NT-pro BNP is ≥ 400 pg/mL

   ii- Is presently in Atrial Fibrillation and NT-pro BNP is ≥ 600 pg/mL

   OR

   B) Patient has had no hospitalization for Heart Failure in the past 9 months AND:

   i- Has had paroxysmal Atrial Fibrillation, is presently in Normal Sinus Rhythm and NT-proBNP is ≥ 600 pg/mL

   ii- Is presently in Atrial Fibrillation and NT-proBNP is ≥ 900 pg/mL

   *Heart Failure Admission is defined as admission to hospital > 24 hours and received treatment for Heart failure
5. Suitable candidate for catheter ablation or rate control therapy for the treatment of AF
6. Age ≥18

Exclusion Criteria:

1. Have an LA dimension > 55 mm as determined by an echocardiography within the previous year
2. Had an acute coronary syndrome or coronary artery bypass surgery within 12 weeks
3. Have rheumatic heart disease, severe aortic or mitral valvular heart disease using the AHA/ACC guidelines
4. Have congenital heart disease including previous ASD repair, persistent left superior vena cava
5. Had prior surgical or percutaneous AF ablation procedure or atrioventricular nodal (AVN) ablation
6. Have a medical condition likely to limit survival to < 1 year
7. Have New York Heart Association (NYHA) class IV heart failure symptoms
8. Have contraindication to systematic anticoagulation
9. Have renal failure requiring dialysis
10. AF due to reversible cause e.g. hyperthyroid state
11. Are pregnant
12. Are included in other clinical trials that will affect the objectives of this study
13. Have a history of non-compliance to medical therapy
14. Are unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 411 (Actual)
Dates: Start 2011-09; Primary Completion 2021-05 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Composite of all-cause mortality and heart failure events | Baseline to a minimum of 24 months
  Heart failure event defined as an admission to a healthcare facility for > 24 hours or clinically significant worsening heart failure leading to an intervention (defined as treatment in an emergency department, a same-day access clinic, or an infusion centre) or unscheduled visits to a healthcare provider for administration of an intravenous diuretic as accepted by FDA and an increase in chronic heart failure therapy

SECONDARY OUTCOMES:
All-cause mortality | Baseline to a minimum of 24 months
  All-cause mortality
Heart Failure events | Baseline to a minimum of 24 months
  Heart failure event defined as an admission to a healthcare facility for > 24 hours or clinically significant worsening heart failure leading to an intervention (defined as treatment in an emergency department, a same-day access clinic, or an infusion centre) or unscheduled visits to a healthcare provider for administration of an intravenous diuretic as accepted by FDA and an increase in chronic heart failure therapy
Health related QoL | Baseline to a minimum of 24 months
  Minnesota Living with Heart Failure. Scoring: The higher the score, the worse the HRQL
Health related QoL | Baseline to a minimum of 24 months
  EuroQol- 5 Dimension. Scoring 0 = worst to 100 = best
Health related QoL | Baseline to a minimum of 24 months
  Atrial Fibrillation Effect on Quality-of-life. Scoring 0 = worst to 100 = best
Exercise capacity | Baseline to a minimum of 24 months
  as determined by 6 Minute Hall walk distance
NT-proBNP/BNP at 1 year and at 2 year follow-up | Baseline to a minimum of 24 months
  NT-proBNP/BNP
All-cause mortality and heart failure events in patients with HF, impaired (LVEF≤45%) LV function and high burden AF | Baseline to a minimum of 24 months
All-cause mortality and heart failure events in patients with HF, preserved (LVEF > 45%) LV function and high burden AF | Baseline to a minimum of 24 months
Health economics | Baseline to a minimum of 24 months
  Cost economics

OTHER OUTCOMES:
LV function and remodeling (LVESVi) at 1 year and 2 year follow-up | Baseline to a minimum of 24 months
  Echocardiogram measure LVESVi
AF Burden at 1 year and 2 year follow-up | Baseline to a minimum of 24 months
  14 Day Continuous ECG monitoring
Total number of heart failure events | Baseline to a minimum of 24 months
  Heart failure event defined as an admission to a healthcare facility for > 24 hours or clinically significant worsening heart failure leading to an intervention (defined as treatment in an emergency department, a same-day access clinic, or an infusion centre) or unscheduled visits to a healthcare provider for administration of an intravenous diuretic as accepted by FDA and an increase in chronic heart failure therapy
Total number of Cardiovascular hospitalizations | Baseline to a minimum of 24 months
  Cardiovascular hospitalizations
Safety (Adverse Events) | Baseline to a minimum of 24 months
  Thromboembolic events, symptomatic Pulmonary vein stenosis, atrio-esophageal fistula, pericardial effusion requiring pericardiocentesis, major bleeding requiring blood transfusion, amiodarone induced thyroid, pulmonary and other toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Tang, MD FRCPC, Principal Investigator — Western University; George Wells, PhD, Principal Investigator — Ottawa Heart Institute Research Corporation
Locations (21):
- Instituto de Cardiologia-FUC RS, Porto Alegre, Rio Grande do Sul, Brazil
- Canada (18):
  - Libin Cardiovascular Institute of Alberta, Calgary, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Vancouver General, Vancouver, British Columbia
  - Royal Jubilee Hospital, Victoria, British Columbia
  - Queen Elizabeth II Health Science, Halifax, Nova Scotia
  - Hamilton Health Sciences Centre, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - St. Mary's General Hospital, Kitchener, Ontario
  - London Health Sciences Centre, London, Ontario
  - Southlake Regional Health Care, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto General Hospital, University Health Network, Toronto, Ontario
  - Institute de Cardiologie de Montréal, Montreal, Quebec
  - CHUM Centre hospitalier universitaire de Montréal, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Insitut universitaire de cardiologie and pneumologie de Quebec, Québec, Quebec
  - CHUS Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec
- Karolinska University Hospital, Stockholm, Sweden
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Parkash R, Wells GA, Rouleau J, Talajic M, Essebag V, Skanes A, Wilton SB, Verma A, Healey JS, Sterns L, Bennett M, Roux JF, Rivard L, Leong-Sit P, Jensen-Urstad M, Jolly U, Philippon F, Sapp JL, Tang ASL. Randomized Ablation-Based Rhythm-Control Versus Rate-Control Trial in Patients With Heart Failure and Atrial Fibrillation: Results from the RAFT-AF trial. Circulation. 2022 Jun 7;145(23):1693-1704. doi: 10.1161/CIRCULATIONAHA.121.057095. Epub 2022 Mar 22. PMID 35313733